CLINICAL TRIAL: NCT01850069
Title: The Use of Near Infrared Spectroscopy (NIRS) to Estimate Intracranial Pressure (ICP)
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Bhiken I. Naik, MD, Assistant Professor, Anesthesiology, University of Virginia
Other Study IDs: 16714
Record Dates: First submitted 2013-04-25; First posted 2013-05-09 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Intracranial Hypertension
Keywords: Intracranial hypertension; intracranial elastance
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intracranial hypertension: Patients with raised intracranial pressure

SUMMARY:
The aim of this study is to determine whether we can predict the intracranial pressure using near infra-red spectroscopy

DETAILED DESCRIPTION:
The management of intracranial hypertension requires the presence of an intracranial pressure monitor. We are investigating whether the waveforms obtained from a near infrared spectroscopy device can predict what the intracranial pressure is non-invasively.

* Patients with intracranial hypertension who are intubated and ventilated in the ICU will be recruited
* we will record there intracranial pressure and systemic arterial pressure
* recordings from the near infrared device will be recorded and analysed off-line
* we will correlate the waveform tracings from near infrared spectroscopy and the arterial tracing

ELIGIBILITY:
Inclusion Criteria:

Patients with an intracranial pressure monitor and arterial catheter who are admitted to the ICU

Exclusion Criteria:

Less than 18 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the ICU with intracranial hypertension, being monitored with an arterial catheter and intraranial pressure monitor
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-01-10 (Actual)

PRIMARY OUTCOMES:
Intracranial elastance | Participants will be followed while an arterial line and intracranial pressure monitor is present duing the ICU admission. This is expected to be an average of 5 days.
  Intracranial elastance (δP/δV)will be measured by dividing the pulse pressure of an invasive arterial blood pressure by the amplitude of high frequency oscillations in the near infrared (NIR) absorbance waveforms.

CONTACTS AND LOCATIONS:
Overall Officials: Bhiken Naik, MBBCh, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brain Trauma Foundation; American Association of Neurological Surgeons; Congress of Neurological Surgeons; Joint Section on Neurotrauma and Critical Care, AANS/CNS; Carney NA. Guidelines for the management of severe traumatic brain injury. Methods. J Neurotrauma. 2007;24 Suppl 1:S3-6. doi: 10.1089/neu.2007.9996. No abstract available. PMID 17511542
- [Background] Rosenberg JB, Shiloh AL, Savel RH, Eisen LA. Non-invasive methods of estimating intracranial pressure. Neurocrit Care. 2011 Dec;15(3):599-608. doi: 10.1007/s12028-011-9545-4. PMID 21519957
- [Background] Lee JK, Kibler KK, Benni PB, Easley RB, Czosnyka M, Smielewski P, Koehler RC, Shaffner DH, Brady KM. Cerebrovascular reactivity measured by near-infrared spectroscopy. Stroke. 2009 May;40(5):1820-6. doi: 10.1161/STROKEAHA.108.536094. Epub 2009 Mar 12. PMID 19286593